CLINICAL TRIAL: NCT06241261
Title: Randomised Clinical Trial to Arrest Early Childhood Caries With a Silver Diamine Fluoride Gel
Brief Title: Arresting Early Childhood Caries With a Silver Diamine Fluoride Gel
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 23-064
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Early Childhood Caries
Keywords: Silver Diamine Fluoride; Caries; Arrest; Gel; Children
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver diamine fluoride gel (Experimental): 38% silver diamine fluoride gel
  Interventions: Drug: Silver diamine fluoride gel
- Silver diamine fluoride solution (Active Comparator): 38% silver diamine fluoride solution
  Interventions: Drug: Silver diamine fluoride solution

INTERVENTIONS:
Drug: Silver diamine fluoride gel — Application of 38% SDF gel every 6 months
  Other Names: SDF gel
  Arms: Silver diamine fluoride gel
Drug: Silver diamine fluoride solution — Application of 38% SDF solution every 6 months
  Other Names: SDF solution
  Arms: Silver diamine fluoride solution

SUMMARY:
The objective is to determine whether the efficacy of a 38% silver diamine fluoride (SDF) gel is non-inferior to a 38% SDF solution for arresting carious lesions in preschool children when applied at half-yearly intervals over a 30-month period.

DETAILED DESCRIPTION:
Aim: Silver diamine fluoride (SDF) is typically available as a 38% aqueous solution, which is runny and difficult to apply. A 38% SDF gel has been introduced but it has not been tested clinically. The objective is to determine whether the efficacy of a 38% SDF gel is non-inferior to a 38% SDF solution for arresting carious lesions in preschool children.

Methods / Design: This non-inferiority randomised clinical trial will recruit 630 3- to 4-year-old children to receive either SDF gel or SDF solution on their carious lesions every 6 months. The primary outcome is the proportion of active carious tooth surfaces that arrest at the 30-month follow-up. The same examiner will conduct all examinations at the kindergartens over 30 months. The examiner, the children, and the children's parents will be blinded to treatments. The parents will be surveyed on their child's oral health-related behaviours and socioeconomic background to allow adjustment for effect modification.

Significance: If the result is as anticipated, SDF gel will prolong contact of SDF with the carious lesion to promote remineralisation. As SDF gel is cost-effective, simple, non-invasive, and non-aerosol-generating, it can be widely recommended for caries control.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy, have at least one tooth with cavitated dentine carious lesion

Exclusion Criteria:

* uncooperative and difficult to manage, with severe forms of hypoplasia of fluorosis or other oral diseases, wearing orthodontic devices or under dental treatment, have major systemic diseases, or are on long-term medication

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 630 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The hardness of cavity on tooth by probing | The follow-up oral examinations will be conducted every 6 months for 30 months totally
  The number of active carious tooth surfaces that become arrested per child

CONTACTS AND LOCATIONS:
Overall Officials: Chun Hung Chu, Ph.D, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng AY, Chen J, Zheng FM, Duangthip D, Chu CH. Arresting Early Childhood Caries with Silver Diamine Fluoride Gel Among Preschool Children: Protocol for a Randomised Clinical Trial. Dent J (Basel). 2024 Dec 22;12(12):419. doi: 10.3390/dj12120419. PMID 39727476